CLINICAL TRIAL: NCT05129566
Title: Comparative Evaluation of Long-term Axial Stability of Two Different Models of Intraocular Lenses in Patients With an Eye Length More Than 26 mm
Brief Title: Evaluation of Axial Stability of Two Models of Intraocular Lenses in Patients With an Eye Length More Than 26 mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Boris Malyugin, Principal Investigator, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #108.1_06092021
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cataract Senile; Myopia, High-Grade; Corneal Astigmatism
Keywords: Axial stability, cataract surgery, IOL, high myopia
MeSH Terms: conditions — Myopia; Astigmatism; Intraocular Lymphoma

STUDY DESIGN:
Intervention Model Description: The first group of patients will receive the IOL Clareon AutonoMe (Alcon, USA), and the second group of patients will receive the IOL Hoya iSert 251 (Japan), 39 eyes in each group, total 78 patients, 78 eyes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL Clareon AutonoMe (Experimental): The first group of patients (39 eyes) who received the monofocal IOL Clareon AutonoMe after the phacoemulsification of cataract.
  Interventions: Procedure: IOL Clareon AutonoMe
- IOL Hoya iSert 251 (Active Comparator): the second group of patients (39 eyes) who received the monofocal IOL Hoya iSert 251 after the phacoemulsification of cataract
  Interventions: Procedure: IOL Hoya iSert 251

INTERVENTIONS:
Procedure: IOL Clareon AutonoMe — Phacoemulsification of cataract with implantation of two types of IOLs - Clareon AutonoMe and Hoya iSert 251. Operations will be performed by one surgeon using the Centurion vision system under control of the Verion navigation system. The Verion system will be used for capsulorhexis and IOL centration (limbus centration).
  Arms: IOL Clareon AutonoMe
Procedure: IOL Hoya iSert 251 — Phacoemulsification of cataract with implantation of two types of IOLs - Clareon AutonoMe and Hoya iSert 251. Operations will be performed by one surgeon using the Centurion vision system under control of the Verion navigation system. The Verion system will be used for capsulorhexis and IOL centration (limbus centration).
  Arms: IOL Hoya iSert 251

SUMMARY:
Some parameters, such as a change in the optic tilt and axial decentration, can affect the optical characteristics of intraocular lenses (IOLs) in postoperative period, which leads to residual refractive errors and other complications.

The stability of the intraocular lens in the eye is largely dependent on the mechanical design of its haptic support elements. Thus, the new Clareon IOL has a flat haptic with a flexible design that minimizes axial changes and allows the IOL to maintain a stable position in a given plane during compression.

Currently there is no published data of the stability for Clareon AutonoMe IOL for long eyes.

The purpose of the current study is to evaluate and compare the axis displacement and stability of optical tilt, visual and refractive results in patients after implantation of two different models of intraocular lenses: Clareon AutonoMe (Alcon, USA) and Hoya iSert 251 (Japan) in the long-term postoperative period (after cataract surgery).

DETAILED DESCRIPTION:
The optical performance of intraocular lenses (IOLs) can be affected by changes in optic tilt and decentration that occur after implantation, resulting in residual refractive errors and other complications. Intraocular lens stability is largely dependent on the mechanical design of the haptics. Clareon IOL has a flat haptic with a flexible design that minimizes axial changes and allows the IOL to maintain a stable position in a given plane during compression.

Based on our knowledge, nobody has compared Clareon AutonoMe and Hoya iSert 251 IOLs in clinical setting.

Scientific Rationale:

This study investigates the stability of IOLs in patients with long axial length. IOL stability on long eyes has a limited clinical data, no in Vivo research has been done. It is known that eyes with long axial length have a large capsule bag. With such eyes, it is difficult to predict the effective lens position.

Each 0,5 mm axial displacement lead to approximately 0,5 D of the refractive error.

For long eyes, it is important to use the latest generation of multi-component IOL calculation formulas for accurately prediction of effective lens position.

The mail purpose of the study is to evaluate and compare the axis displacement and stability of optical tilt, visual and refractive results in patients after implantation of two different models of intraocular lenses: Clareon AutonoMe (Alcon, USA) and Hoya iSert 251 (Japan) in the long-term postoperative period (after cataract surgery).

The research purpose is to evaluate the prediction error for each IOL calculation formula (Barrett Universal II, Kane, EVO, Holladay I with Van Koch correction)

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 50 years and older with indicated cataract surgery.
* Signed informed consent, given by the participant or his/her legal representative.
* Ability to understand Russian spoken and written language.
* Sanitated oral cavity.
* Intraocular pressure in normal range.
* Axial eye length> 26 mm.
* Corneal astigmatism <1.0 diopters.
* The presence of age-related cataract with high myopia and low visual acuity (less than 0.5 with correction), the cornea thickness in the central optical zone is not less than 500 microns and not more than 600 microns, and the density of endothelial cells is higher than 2300 cells / mm2.
* Patients who have passed the entire tests for hospitalization in hospital and also have received the admission (the conclusion) of the therapist for the surgery.

Exclusion Criteria:

* Inability to give signed informed consent.
* Age under 50 years.
* History of allergic reactions to antibiotics, glucocorticosteroids, medications for local and general anesthesia.
* Diagnosed neoplastic process or treatment for tumor disease.
* Positive tests for infectious: HIV, syphilis, Hepatitis B, Hepatitis C.
* Any medical, psychiatric and/or condition, including cachexia, or social conditions that the investigator believes would interfere with or contraindicate adherence to the research protocol or the ability to provide signed informed consent.
* Active ophthalmic infection.
* Uncontrolled glaucoma
* Retinal defunctioning (no light perception and/or retinal detachment).
* Absence of the electric activity of the optic nerve and/or retina.
* Concomitant ocular pathology, such as the subluxation of the lens, glaucoma, pathology of the central retina, diabetic retinopathy, scars and opacities of the cornea, keratoconus, pathology of the corneal endothelium (Fuchs corneal dystrophy), pseudoexfoliative syndrome with pronounced impairment of the diaphragmatic function of the pupil, a non-functioning retina (lack of light perception and/or its detachment according to ultrasound examination), lack of electrical activity of the optic nerve and retina according to electrophysiological examination, etc.
* Patients with a serious general medical condition.
* Systemic use / administration of drugs that may affect the anatomical or functional characteristics of the cornea (amiodarone, β-blockers, tetracycline, etc.)
* Any pathology of the eye associated with myopia and myopic changes inside the eye (for example, myopic staphyloma) that may affect the results of the study.
* Regular intake of medications that may affect the proper function of the eye (antiglaucoma drugs, antibiotics, systemic immunosuppressive therapy, etc.)
* Systemic pathologies with possible damage to the cornea.
* Amblyopia.
* Any other concomitant ocular pathology, trauma or surgery in history.
* A patient who cannot adhere to the schedule of visits for research or treatment (for example, patients from other cities).
* Suspected drug or alcohol abuse.

Ages: 50 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Intraocular lens axial displacement | 6 months
  Axial displacement of the intraocular lens, stable position of the intraocular lens in the capsule bag after surgery, optics tilt, deviation from baseline, the distance from the corneal epithelium to the anterior surface of the intraocular lens, the stretching degree of the surgical wound will be assessed by the anterior segment OCT (AS-OCT).

SECONDARY OUTCOMES:
Near and distance vision visual acuity | 6 months
  Improving the clarity of images of observed objects. For one focus distance (reading and working at near / far (depending on the calculation of the IOL for emmetropia or weak myopic refraction) / intermediate distance, it is possible to use spectacle correction in the postoperative period.
Patient's subjective satisfaction of with the quality of vision | 6 months
  Increased subjective satisfaction of patients with the quality of vision after surgery will be assessed using the VF-14 questionnaire (Steinberg E.P., 1994).
Deviation from emmetropic refraction | 6 months
  Accurate IOL calculation before surgery.
Number of intra- and postoperative complications | 6 months
  Intra- and postoperative complications in the operated eye will be assessed according to the observation data of the research subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Boris E Malyugin, MD, PhD, Principal Investigator — The S. Fyodorov Eye Microsurgery Federal State Institution
Locations (1):
- The S. N. Fyodorov Eye Microsurgery Federal State Institution, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share Clinical Study Report, present and publish results of the study.
Supporting Information: CSR
Time Frame: During the study and after.
Access Criteria: upon request

REFERENCES:
- [Background] Wirtitsch MG, Findl O, Menapace R, Kriechbaum K, Koeppl C, Buehl W, Drexler W. Effect of haptic design on change in axial lens position after cataract surgery. J Cataract Refract Surg. 2004 Jan;30(1):45-51. doi: 10.1016/S0886-3350(03)00459-0. PMID 14967267
- [Background] Remon L, Cabeza-Gil I, Calvo B, Poyales F, Garzon N. Biomechanical Stability of Three Intraocular Lenses With Different Haptic Designs: In Silico and In Vivo Evaluation. J Refract Surg. 2020 Sep 1;36(9):617-624. doi: 10.3928/1081597X-20200713-02. PMID 32901830
- [Background] Bang S, Edell E, Yu Q, Pratzer K, Stark W. Accuracy of intraocular lens calculations using the IOLMaster in eyes with long axial length and a comparison of various formulas. Ophthalmology. 2011 Mar;118(3):503-6. doi: 10.1016/j.ophtha.2010.07.008. Epub 2010 Sep 29. PMID 20884057
- [Background] Lane S, Collins S, Das KK, Maass S, Thatthamla I, Schatz H, Van Noy S, Jain R. Evaluation of intraocular lens mechanical stability. J Cataract Refract Surg. 2019 Apr;45(4):501-506. doi: 10.1016/j.jcrs.2018.10.043. Epub 2019 Jan 25. PMID 30686704